CLINICAL TRIAL: NCT03442413
Title: The Influence of Nicotinic Hepatic Metabolism on Neuroreceptor Substrates of Nicotine Addiction
Brief Title: Nicotinic Hepatic Metabolism on Neuroreceptor Substrates of Nicotine Addiction
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 828090
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Smoking, Tobacco
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 2-[18F]-FA PET/CT (Experimental): Subjects will participate in two separate 10-hour PET/CT Scan Sessions (each with 2 hours of actual PET/CT scanning): one following an overnight abstinence and one following two overnights of abstinence. To achieve and confirm two overnights of abstinence, participants will present to the inpatient CHPS the day prior to the scheduled scan and stay overnight
  Interventions: Drug: 2-[18F]-FA PET/CT; Drug: I.V. Nicotine

INTERVENTIONS:
Drug: 2-[18F]-FA PET/CT — 2-[18F]FA is a highly specific radiotracer which has been used successfully to image nicotinic acetylcholine receptors in the human brain to characterize the effects of nicotine exposure (via smoking) on these receptors.
Drug: I.V. Nicotine — Subjects in our study will receive intravenous nicotine at the adaptation session and each of the PET scans, close to the amount of nicotine absorbed from smoking 1/10 cigarette.

SUMMARY:
Physically healthy adult smokers may be eligible for this study. Volunteers may participate in this study if they are 18 - 65 years old.

Subjects will participate in two separate 7-hour PET/CT Scan Sessions (each with 2 hours of actual PET/CT scanning): one following an overnight abstinence and one following two overnights of abstinence. To achieve and confirm two overnights of abstinence, participants will present to the inpatient CHPS the day prior to the scheduled scan and stay overnight.

The 2-[18F]-FA PET/CT brain scans will consist of an injection followed by an 7-hour infusion of 2-[18F]-FA. The scan session will begin at approximately 4 hours after the bolus injection. The PET/CT scan will occur in two segments. Starting at approximately 4 hours post bolus and infusion start, we will scan for approximately 90 minutes with a bolus injection of IV nicotine that will occur approximately 15 minutes into the scanning procedure. There will be a break in scanning of approximately 60 minutes, during which subjects will be allowed to get off the scanner and use the restroom, if necessary. The second scan segment will start at approximately 6.5 hours post bolus injection, t. This segment will last approximately 30 minutes. The pre and post nicotine images will be analyzed to evaluate for differences in receptor uptake after the nicotine "challenge".

Subjects will have a structural Brain MRI performed within 1 year prior to study enrollment or subjects who have not had a Brain MRI that is deemed acceptable for use for this study will undergo a research Brain MRI after consent.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be 18-65 years of age
2. Self-reported cigarette smoking history of at least 10 cigarettes/day for at least 6 months prior to enrollment
3. Carbon monoxide reading > 10 ppm at the initial screening session
4. Participants agree to be compliant with all study procedures including smoking abstinence and willingness to complete over-night stays at the Hospital of the University of Pennsylvania
5. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Women who are pregnant at the time of screening will not be eligible for this study. A urine pregnancy test will be performed in women of childbearing potential at screening.
2. Self-reported regular (daily) use of chewing tobacco, snuff or snus
3. Current enrollment in a smoking cessation or research program involving the use of nicotine substitutes
4. History within one year or currently receiving treatment for substance abuse other than nicotine (e,g,, alcohol, opioids, cocaine, marijuana, or stimulants)
5. Current use of cocaine, methamphetamines or other psychoactive substances per self-report and/or positive urine drug screen at the initial screening session
6. Self-reported current alcohol consumption that exceeds greater than 25 drinks per week in men and 18 drinks per week in women
7. BrAC reading greater than or equal to 0.01% at the initial screening session
8. History of kidney and/or liver disease per medical record review or self-reported
9. Uncontrolled hypertension (defined as Systolic BP > 160 and/or Diastolic BP > 100 at the screening intake session)
10. History of Posttraumatic Stress Disorder (PTSD), bipolar disorder, schizophrenia or other psychotic disorder or Attention-Deficit/Hyperactivity Disorder (ADHD) as assessed by medical record review and/or self-report. History of unipolar depression or anxiety disorder may be accepted; current depression or anxiety may be accepted if the severity does not require psychoactive medication as assessed by medical record review and/or self-report.
11. History of head trauma, that in the opinion of an investigator may interfere with the uptake of [18F]2-FA, as assessed by medical record review and/or self-report
12. Current use or recent discontinuation (within the last 14 days) of any of the following:

    1. Smoking cessation medication (e.g. Zyban, Wellbutrin, Wellbutrin SR, Chantix).
    2. Anti-psychotic medications.
    3. Certain medications used to treat depression, including SSRIs, Wellbutrin, MAOIs, and tricyclic antidepressants.
    4. Prescription stimulants (e.g. Provigil, Ritalin, Adderall).
13. Current use of any of the following:

    1. Nicotine replacement therapy (NRT).
    2. Tagamet (cimetidine).
    3. Heart medications such as digoxin, quinidine, nitroglycerin. Use of these medications may result in ineligibility and will therefore be evaluated on a case-by-case basis by the Study Physician.
    4. Anti-coagulants (e.g. Coumadin, Warfarin).
    5. Any drug the investigator determines could interfere with scan results.
14. Daily use of any of the following:

    1. Opiate-containing medications for chronic pain; If a participant reports taking an opiate-containing medication every day for the 14 days prior to the telephone screen and/or the Intake Session, the participant will be ineligible.
    2. Rescue Inhalers (e.g. Albuterol, Proventil, Ventolin, or Maxair).
15. Any contraindication to brain MRI
16. Any current medical condition, psychiatric disorder, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
Duration of abstinence affects brain nAChR availability in smokers | 2 years
  To determine how duration of abstinence affects brain nAChR availability in smokers who metabolize nicotine at slow and normal rates (measured by the nicotine-metabolite ratio (NMR)).
How nicotine administration affects nAChR availability during early abstinence in smokers | 2 years
  To compare how nicotine administration affects nAChR availability during early abstinence in smokers who metabolize nicotine at slow and normal rates (measured by the NMR).

SECONDARY OUTCOMES:
Standard measures of cigarette craving and withdrawal to nAChR availability in smokers | 2 years
  To correlate standard measures of cigarette craving and withdrawal to nAChR availability in smokers who metabolize nicotine at slow and normal rates (measured by the NMR) who are abstinent, before and after administration of IV nicotine

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No